CLINICAL TRIAL: NCT01011673
Title: An RCT of Metoclopramide/Diphenhydramine vs. Ketorolac Alone for Tension-type Headache
Brief Title: Metoclopramide Versus Ketorolac for Tension-type Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-08-249
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Headache
Keywords: headache; tension-type headache
MeSH Terms: conditions — Headache; Tension-Type Headache | interventions — Metoclopramide; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Active Comparator): Ketorolac 30mg IVSS
  Interventions: Drug: Ketorolac
- Metoclopramide (Active Comparator): metoclopramide 20mg IVSS + diphenhydramine 25mg IVSS
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Metoclopramide — metoclopramide 20mg IVSS + diphenhydramine 25mg IVSS
  Other Names: Reglan
  Arms: Metoclopramide
Drug: Ketorolac — ketorolac 30mg IVSS
  Other Names: Toradol
  Arms: Ketorolac

SUMMARY:
Occasionally, episodic tension-type headache may be severe enough to require an emergency department (ED) visit. The purpose of this study is to compare two commonly used medications to see which is better for tension type headache. Patients who present to the ED with an acute tension-type headache requiring treatment with injectable medication will be randomized to metoclopramide or ketorolac.

ELIGIBILITY:
Inclusion Criteria:

* Acute tension type headache

Exclusion Criteria:

* Contraindications to investigational medications
* Secondary cause of headache

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Friedman BW, Adewunmi V, Campbell C, Solorzano C, Esses D, Bijur PE, Gallagher EJ. A randomized trial of intravenous ketorolac versus intravenous metoclopramide plus diphenhydramine for tension-type and all nonmigraine, noncluster recurrent headaches. Ann Emerg Med. 2013 Oct;62(4):311-318.e4. doi: 10.1016/j.annemergmed.2013.03.017. Epub 2013 Apr 6. PMID 23567060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from one emergency department (ED) in the Bronx, NY
Groups:
- Ketorolac: Ketorolac 30 mg, administered intravenously over 15 minutes
- Metoclopramide: metoclopramide 20 mg + diphenhydramine 25 mg, administered intravenously over 15 minutes
Period: Randomized
Arm/Group | Ketorolac | Metoclopramide
Started | 62 | 61
Completed | 60 (2 patients were randomized but not included in analyses bc they did not truly meet study criteria.) | 60 (1 patient was randomized but not included in analyses bc they did not truly meet study criteria.)
Not Completed | 2 | 1
Not completed — Secondary headache | 2 | 1
Period: Emergency Department Portion
Arm/Group | Ketorolac | Metoclopramide
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0
Period: 24 Hour Follow-up
Arm/Group | Ketorolac | Metoclopramide
Started | 60 | 60
Completed | 57 | 57
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Metoclopramide | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 39 (12) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 12 | 18 | 30
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: At baseline at at 60 minutes, all patients were asked to describe their pain on a scale from 0 to 10, with 0 representing no pain and 10 the worst imaginable. The primary outcome is the 60 minute score subtracted from the baseline score
Time Frame: Baseline, 60 minutes
Population: 3 randomized patients were not included in this analysis. During the ED visit, these patients were diagnosed with intracranial hemorrhage, brain abscess, and malaria and therefore did not truly have a primary headache disorder. Including these patients, 123 were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Metoclopramide
Number analyzed (Participants) | 60 | 60
units on a scale | 3.8 (2.6) | 5.1 (2.8)

2. Secondary Outcome: Satisfaction Scores
Description: 24 hours after the emergency department visit, patients were asked, "The next time you come to the Er with this type of headache, do you want to receive the same medication?" Affirmative answers are tabulated here.
Time Frame: 24 hours
Population: 3 patients in each group were lost to follow-up. All others are tabulated here.
Measure: Number; unit: participants
Arm/Group | Ketorolac | Metoclopramide
Number analyzed (Participants) | 57 | 57
participants | 45 | 53

ADVERSE EVENTS:
Arm/Group | Ketorolac | Metoclopramide
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 14/60 | 12/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=60) | Metoclopramide (N=60)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Akathisia (Nervous system disorders) | 8 (8) | 8 (8)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No